CLINICAL TRIAL: NCT01979939
Title: A Phase 3 Evaluation of a Daclatasvir/Asunaprevir/BMS-791325 Fixed Dose Combination in Non-cirrhotic Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: UNITY 1: A Study of an Investigational Treatment Regimen of Daclatasvir (DCV) + Asunaprevir (ASV) + BMS-791325 in a Fixed Dose Combination (the DCV 3DAA (Direct Acting Antiviral) Regimen) for 12 Weeks for the Treatment of Chronic Hepatitis C Virus (HCV) Genotype 1 Infection in Non-cirrhotic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI443-102; 2013-002468-20 (EudraCT Number)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1: DCV/ASV/BMS-791325 in treatment-naive subjects (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325
- A 2: DCV/ASV/BMS-791325 in treatment-experienced subjects (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325

INTERVENTIONS:
Drug: DCV/ASV/BMS-791325

SUMMARY:
To demonstrate the effectiveness of DCV 3DAA fixed dose regimen in treatment naive and treatment experienced non-cirrhotic subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1
* HCV RNA ≥ 10,000 IU/mL at screening
* Treatment-naïve subjects with no previous exposure to an interferon formulation (ie, IFNα, pegIFNα), RBV, or HCV DAA (protease, polymerase inhibitor, etc.)
* Treatment-experienced subjects are eligible

Exclusion Criteria:

* Evidence of cirrhosis
* Liver or any other organ transplant
* Current or known history of cancer within 5 years prior to enrollment
* Documented or suspected HCC
* Evidence of decompensated liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects in the naive cohort with sustained virologic response (SVR) 12 | Post-Treatment Week 12
  SVR12 is defined as HCV ribonucleic acid (RNA) < limit of quantitation (LOQ) target detected or target not detected (LOQ TD/TND) at post treatment Week 12

SECONDARY OUTCOMES:
Proportion of subjects in the experienced cohort with SVR12 | Follow up Week 12
Proportion of subjects in each cohort who achieve HCV RNA <LOQ TD/TND | On-treatment Weeks: 1, 2, 4, 6, 8, and 12; post treatment Weeks 4 (SVR4), 8 (SVR8) and 24 (SVR24)
Proportion of subjects in each cohort who achieve HCV RNA <LOQ TND | On-treatment Weeks: 1, 2, 4, 6, 8, and 12; post treatment weeks 4, 8, 12 and 24
Safety measured by frequency of serious AEs (SAEs) and discontinuations due to adverse events (AEs) through the end of treatment in each cohort | Up to post treatment week 4 (±7 days)
Proportion of anemia defined as Hg <10 g/dL on-treatment and Hg ≥10 g/dL at baseline , in each cohort | Up to post treatment week 4 (±7 days)
Rates of selected grade 3-4 lab abnormalities (hematologic and liver function) in each cohort | Up to post treatment week 4 (±7 days)
Proportion of subjects in each cohort achieving SVR12 associated with HCV geno subtype 1a vs 1b | Post treatment week 12
Proportion of subjects in each cohort achieving SVR12 associated with IL28B rs12979860 single nucleotide polymorphism (SNP) status (CC genotype or non-CC genotype) | Post treatment week 12
Proportion of subjects in each cohort achieving SVR12 associated with stage of liver fibrosis | Post treatment week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (62):
- United States (42):
  - Scripps Clinic, La Jolla, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - University Of Chicago Medical Center, Chicago, Illinois
  - Indiana University Med Center, Indianapolis, Indiana
  - Digestive Disease Associates, P.A., Catonsville, Maryland
  - Johns Hopkins Medical Institutions, Lutherville, Maryland
  - Henry Ford Health System, Novi, Michigan
  - Kansas City Care Clinic, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - The Gastroenterology Group Of South Jersey, Vineland, New Jersey
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Weill Cornell Medical College, New York, New York
  - Premier Medical Group Of The Hudson Valley, Pc, Poughkeepsie, New York
  - James J Peters Vamc, The Bronx, New York
  - Asheville Gastroenterology Associates, Pa, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Trial Management Associates, Llc, Wilmington, North Carolina
  - Digestive Health Specialists, Pa, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center, Ctr For Liver Diseases, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Quality Medical Research Pllc, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor St. Luke'S Medical Center, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Mt Vernon Endoscopy Center, Alexandria, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours St. Mary'S Hospital Of Richmond, Inc., Newport News, Virginia
  - Digestive And Liver Disease Specialists, Norfolk, Virginia
  - Dean Clinic, Madison, Wisconsin
- Australia (7):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Clayton
- Canada (6):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- France (6):
  - Local Institution, Clichy
  - Local Institution, Limoges
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Vandœuvre-lès-Nancy
- Fundacion De Investigacion De Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Poordad F, Sievert W, Mollison L, Bennett M, Tse E, Brau N, Levin J, Sepe T, Lee SS, Angus P, Conway B, Pol S, Boyer N, Bronowicki JP, Jacobson I, Muir AJ, Reddy KR, Tam E, Ortiz-Lasanta G, de Ledinghen V, Sulkowski M, Boparai N, McPhee F, Hughes E, Swenson ES, Yin PD; UNITY-1 Study Group. Fixed-dose combination therapy with daclatasvir, asunaprevir, and beclabuvir for noncirrhotic patients with HCV genotype 1 infection. JAMA. 2015 May 5;313(17):1728-35. doi: 10.1001/jama.2015.3860. PMID 25942723
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx